CLINICAL TRIAL: NCT01857076
Title: Surgical Treatment in Diabetic Patients With Grade 1 Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Sirio-Libanes (Other)
Responsible Party: Principal Investigator, Cláudia Cozer, Md, Hospital Sirio-Libanes
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSL 2012-01; HSL 2012-01 (Other: CEPesq Register Number); 00747112.3.0000.5461 (Registry Identifier: CAAE)
Record Dates: First submitted 2013-05-07; First posted 2013-05-20 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2013-05

CONDITIONS: Obesity; Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes mellitus; Grade I obesity; Inadequate glycemic control
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Clinical (Active Comparator): Subject submitted to clinical obesity treatment
  Interventions: Other: Clinical
- Gastric bypass surgery (Active Comparator): Subjects submitted to Gastric Bypass Surgery
  Interventions: Procedure: Gastric bypass surgery
- Surgical ileal transposition with sleeve (Active Comparator): Subjects submitted to surgical ileal transposition with sleeve
  Interventions: Procedure: Surgical ileal transposition with sleeve

INTERVENTIONS:
Procedure: Gastric bypass surgery — Gastric bypass surgery performed laparoscopically
  Arms: Gastric bypass surgery
Procedure: Surgical ileal transposition with sleeve — Surgical Treatment with Ileal Transposition in the duodenum and Vertical Sleeve Gastrectomy through laparoscopic surgery.
  Arms: Surgical ileal transposition with sleeve
Other: Clinical — The study subjects allocated for clinical treatment will have these treatment divided into three phases. The first one based on glycemic control through weight loss, the second one based on anti-hyperglycemic medications and the last one based on medical monitoring for a further twelve months for the maintenance of the results.
  Arms: Clinical

SUMMARY:
There will be a randomized clinical trial, non-blind, 3-arm treatment (medical, surgical, gastric bypass and ileal transposition surgery with and sleeve), which will be conducted in a single center - S.B.S. Hospital Sirio Libanês, including 75 research subjects with type 2 diabetes mellitus and obesity class I. In order to compare the effect of weight loss on glycemic control among medical and surgical groups, and after 2 years of follow up, the results of efficacy, safety and maintenance will be compared between the three groups.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman with Type 2 diabetes mellitus (DM) aged between 25 and 65 years, with time since diagnosis of diabetes less than 10 years.
* Grade I obesity (BMI between 30-35)
* Inadequate glycemic control with HbA1c between 7.0 to 9.5% at baseline, in the presence of drug treatment for diabetes in the last year.
* Reserve pancreatic C-peptide> 1.0 at baseline.
* Overweight stable defined as BMI> 30 in the last two years.

Exclusion Criteria:

* History ketoacidosis, diabetes mellitus type 1, diabetes followed by pancreatitis.
* Repetition of measurements (ie, 2 or more within 1 week) fasting plasma glucose(FPG) > 240 mg / dL during the pre-treatment.
* History of Severe Proliferative Diabetic Retinopathy.
* Autonomic neuropathy.
* Loss or gain significant weight within the last 12 weeks (range, 5% body weight)
* Renal insufficiency
* History of renal disease treated with immunosuppressive therapy, history of dialysis or kidney transplantation.
* Presence of other renal diseases (eg nephrotic syndrome, glomerulonephritis)
* Acute myocardial infarction, unstable angina (NYHA class III-IV), revascularization or stroke within the previous 3 months of the initial visit.
* Uncontrolled hypertension defined as diastolic blood pressure> 100mm/Hg and diastolic blood pressure> 160mm/Hg at the initial visit.
* History of Hepatitis B or Hepatitis C.
* Criteria for Hepatic insufficiency defined as Child B and C liver disease clinically active and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) above 3 times the upper limit of normal.
* History of prior bariatric surgery.
* Inflammatory Bowel Disease.
* History neoplasm within the last 5 years (except for squamous cell carcinoma and basal skin and cervical carcinoma in situ)
* Clinically important hematologic disorder (symptomatic anemia, bone marrow proliferative disorders, thrombocytopenia, ..)
* History antibody positive human immunodeficiency virus (HIV)
* Surgery with general anesthesia within 12 weeks prior to the initial visit or incomplete recovery from prior surgery.
* History of drug or alcohol abuse within 3 years before the initial visit.
* Pregnancy or breastfeeding or planning pregnancy in the next two years.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2013-02; Primary Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Glycemic blood rates | In 2 years
  Comparison of efficacy and safety in glycemic control between the medical and surgical treatment.
Glycemic blood rates | In 2 years
  Comparison of efficacy and safety in glycemic control between the two surgical modalities.
Diabetes remission evaluated by patients glycemic rates | In 2 years
  Comparison of diabetes remission between the two surgical modalities.

SECONDARY OUTCOMES:
Weight loss | In 2 years.
  Comparison of efficacy in the control of overweight in the medical and surgical treatment.
Decrease in blood lipid | In 2 years
  Comparison of the effectiveness in controlling lipid between the medical and surgical treatment.
Quality of life evaluation | In 2 years
  Comparison of quality of life between the medical and surgical treatment through specific interviews
Number of Early Adverse Events | In 2 years
  Comparison of early complications between the two surgical modalities.
Number os Nutricional Complications | In 2 years
  Comparison of nutritional complications between the two surgical modalities.
Number of Late Adverse Events | In 2 years
  Comparison of late complications between the two surgical modalities.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Cozer, Md, Principal Investigator — Hospital Sírio-Libanês
Locations (1):
- Hospital Sírio Libanês Teaching and Research Center, São Paulo, São Paulo, Brazil